CLINICAL TRIAL: NCT05822232
Title: A Randomized Controlled Trial Comparing the FreeStyle Libre 2 Continuous Glucose Monitoring vs Point of Care Glucose Testing for the Management of Subjects With Type 2 Diabetes After Hospital Discharge: FreeStyle Libre 2 Discharge Trial
Brief Title: FreeStyle Libre 2 Discharge Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: Abbott Diabetes Care (Industry); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022.050-2
Record Dates: First submitted 2022-12-01; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemia
Keywords: Hospital discharge; algorithm; CGM; technology; type 2 diabetes; hospital hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FreeStyle Libre 2 (Active Comparator): Subjects randomized to Group 1: FreeStyle Libre 2 will wear two FreeStyle Libre CGM sensors for 12-14 days three times over a 12-week (3 month) period. They will have two sensors inserted under their skin:
  FreeStyle Libre 2 sensor with display on, meaning they will be able to see their blood sugar values on the mobile application or a reader.
  FreeStyle Libre Pro sensor is used without mobile application or reader. This sensor is place as a backup in case the information is missing from the Libre 2 sensor.
  Interventions: Device: FreeStyle Libre 2 CGM; Device: FreeStyle Libre Pro blinded CGM
- Point of Care (POC) Self-Monitoring of Blood Glucose (SMBG) testing (Active Comparator): Subjects randomized to Group 2: Point of Care (POC) Self-Monitoring of Blood Glucose (SMBG) testing will wear one FreeStyle Libre Pro CGM sensor without using the mobile application or reader (blinded). These subjects will have the one sensor inserted under their skin but you will not see sugar values on the CGM. Subjects will wear the CGM for 12-14 days three times over a 12-week (3 month) period but will not use the CGM to monitor and control their blood sugar. Instead, they will monitor their sugar values by the standard method of fingerstick before each meal and at bedtime.
  Interventions: Device: FreeStyle Libre Pro blinded CGM; Device: FreeStyle Precision Neo blood glucose meter

INTERVENTIONS:
Device: FreeStyle Libre 2 CGM — FreeStyle Libre 2 CGM is FDA-approved and will be used according to FDA-approved labeling
  Arms: FreeStyle Libre 2
Device: FreeStyle Libre Pro blinded CGM — FreeStyle Libre Pro blinded CGM is FDA-approved and will be used according to FDA-approved labeling
Device: FreeStyle Precision Neo blood glucose meter — FreeStyle Precision Neo blood glucose meter is FDA-approved and will be used according to FDA-approved labeling
  Arms: Point of Care (POC) Self-Monitoring of Blood Glucose (SMBG) testing

SUMMARY:
The goal of this clinical trial is to learn about the benefits of using aa Continuous Glucose Monitoring (CGM) system in patients with diabetes following discharge from the hospital. The main question it aims to answer is:

• If the use of CGM with alarms is safe and effective for managing low and/or high blood sugars when compared with performing finger sticks several times per day

Participants will wear one or two FreeStyle Libre CGM sensors for 12-14 days three times over a 12-week (3 month) period. This means that they will have the one to two sensors inserted under their skin. They will be asked to come to the study site four times and complete two phone calls with research staff over the 12-week period.

Researchers will compare the LibreView CGM group to the Standard of Care group to see if the use of continuous glucose monitoring (CGM) reduces risk of low blood sugar in patients with type 2 diabetes (T2D) after hospital discharge when compared with the current standard method.

DETAILED DESCRIPTION:
The purpose of this study is to look at the benefits of using Continuous Glucose Monitoring (CGM) system for patients with diabetes following discharge from the hospital. CGM devices measure blood sugar every few minutes using a sensor inserted under the skin.

In this study, we will compare the CGM method to the current usual (standard-of-care) method, which involves taking blood samples by fingerstick before meals and at bedtime. The CGM system recognizes low and high blood sugars throughout the day and night. The CGM system used in this study also has an alarm feature that alerts the user if blood sugar levels are too high or too low. In this study we will test if the use of CGM with alarms is safe and effective for managing low and/or high blood sugars when compared with performing finger sticks several times per day, which some diabetes patients find painful and burdensome.

In this study, 50% of participants will use the CGM method and 50% will use the fingerstick method to measure and control their glucose. The researchers will compare the two groups to answer the question if the use of continuous glucose monitoring (CGM) reduces risk of low blood sugar in patients with type 2 diabetes (T2D) after hospital discharge when compared with the current standard method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females ≥18 years of age admitted to general medicine and surgery services.
* 2. Known history of T2D treated with oral antidiabetic agents (sulfonylureas, meglitinides, alpha-glucosidase inhibitors, thiazolidinedione, DPP-4 inhibitors, SGLT2- inhibitors), GLP1-RAs (exenatide, liraglutide, dulaglutide, semaglutide) or insulin therapy (human regular or rapid-acting analogs or ultra-rapid analogs [ lispro, aspart, glulisine, fast acting insulin aspart, insulin lispro]), intermediate acting (NPH and premixed formulations) or long-acting basal (glargine, detemir, degludec) formulations.
* 3. Discharged on insulin therapy consisting of basal therapy 1) with or without bolus insulin and also 2) with or without other diabetes drugs.

Exclusion Criteria:

* 1. Subjects admitted with a diagnosis of diabetic ketoacidosis or hyperosmolar hyperglycemic state.
* 2. Subjects using CGM technology prior to admission
* 3. Subjects with type 1 diabetes
* 4. Subjects not willing to receive insulin injections or test POC 4 times daily
* 5. Subjects discharged from the hospital on diabetes therapy that does not include basal insulin.
* 6. Subjects not willing to wear a CGM device
* 7. Pregnant women
* 8. Subjects with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension) and end-stage kidney disease (eGFR< 30 ml/min), dialysis, critically ill or terminal illness.
* 9. Subjects with history of cognitive impairment, dementia, or mental condition rendering the subject unable to understand the nature and consequences of the study.
* 10. Subjects expected to be readmitted to the hospital within 3 months post-discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | 2 weeks
  Frequency of overall and nocturnal hypoglycemia (< 70 mg/dl) by capillary POC testing and by FreeStyle Libre 2 CGM
Safety Endpoint | 4 weeks
  Frequency of overall and nocturnal hypoglycemia (< 70 mg/dl) by capillary POC testing and by FreeStyle Libre 2 CGM
Safety Endpoint | 12 weeks
  Frequency of overall and nocturnal hypoglycemia (< 70 mg/dl) by capillary POC testing and by FreeStyle Libre 2 CGM
Efficacy endpoint | 2 weeks
  Glycemic control, as measured by mean daily glucose concentration between groups by capillary POC testing and by CGM
Efficacy endpoint | 4 weeks
  Glycemic control, as measured by mean daily glucose concentration between groups by capillary POC testing and by CGM
Efficacy endpoint | 12 weeks
  Glycemic control, as measured by mean daily glucose concentration between groups by capillary POC testing and by CGM

CONTACTS AND LOCATIONS:
Overall Officials: David Klonoff, MD, Principal Investigator — Sutter Health, Diabetes Research Institute
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Division of Endocrinology, Department of Medicine, Emory University School of Medicine, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No